CLINICAL TRIAL: NCT04326582
Title: Arthritis in Assiut University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Masoud Adb-Elmonem, Principal Investigator of pediatrics, Assiut University
Other Study IDs: Arthiritis in children
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — Determine of percentage of each type of arthritis in children, it's prognosis and outcome of treatment in comparison with international guidelines

SUMMARY:
* To define prevalence of different types of arthritis in patients attending Assiut University Children Hospital (AUCH)
* To define prognosis of these different types
* To evaluate management of arthritis in Assiut University Children Hospital, in comparison to international guidelines

DETAILED DESCRIPTION:
Arthritis is defined as inflammation of the joint, Patients have symptoms of joint pain, stiffness, swelling, redness, warmth and decreased range of motion of the affected joints. Arthritis may be caused by transient synovitis, juvenile idiopathic arthritis ( JIA), reactive arthritis, viral arthritis and other inflammatory diseases; septic arthritis also occurs as a complication of bacteraemia in children. The overall incidence of arthritis and its causes are not well documented in children, and have even been reported to be unknown.Two population-based studies have described the incidence of different diagnoses of arthritis in childhood. Both of these studies were performed in Northern Europe and reported that transient synovitis is the most common cause.

The outcome and treatment of arthritis depend on its etiology. Children with transient synovitis do not need any surgical procedures and are treated symptomatically at home. However, children with septic arthritis require early diagnosis and hospital treatment, including surgical joint drainage and intravenous antibiotics so that septicaemia and joint damage can be avoided.

JIA is one of the more common chronic diseases of childhood with a prevalence of approximately 1 per 1,000 .

Criteria and classification Three groups have developed sets of criteria to classify children with arthritis: The American College of Rheumatology (ACR), The European League Against Rheumatism (EULAR), and The International League of Associations for Rheumatology (ILAR).

* THE ILAR classification of JIA includes the following categories:
* systemic-onset JIA
* persistent or extended oligoarthritis
* Rheumatoid factor (RF)-positive polyarthritis
* RF-negative polyarthritis
* Psoriatic JIA
* Undifferentiated(disease does not meet criteria for any of the other subgroups, or it meets more than 1 criterion)

  * Septic arthritis was defined as arthritis associated with bacteria isolated from blood or synovial fluid.
  * Arthritis that did not retrospectively fulfil criteria for septic arthritis, JIA or other well-established diagnoses (haemarthrosis, Kawasaki disease, malignant disease, Gaucher disease, systemic lupus erythematosus, villo-nodular synovitis, dermatomyositis and chronic recurrent multifocal osteitis) was classified as 'arthritis without any definitive diagnosis.
* Although acute monoarthritis (as for instance septic arthritis) is usually considered to be a medical emergency, it is not often realized that patients with polyarthritis also need to be evaluated promptly to ensure timely management. Delays in diagnosis and/or treatment may result in significant morbidity, as for example in rheumatic fever and Kawasaki disease. It cannot be overemphasized enough that the most important clues to underlying etiology in a patient with polyarticular disease are found not in the investigations but in the clinical history and physical examination. Some investigations (e.g. radiographs of joints) are commonly done but may have little or no role in the initial assessment of the patient. Polyarticular joint disease has multi-factorial etiology. It may present acutely as in self limiting viral illnesses or it can be the beginning of a chronic sinister disease. The underlying etiological process can be infectious or post infectious, a rheumatological disease or a manifestation of systemic disease. The disease may evolve over days or sometimes weeks, thereby making the diagnosis difficult at the time of presentation. Viral infections (for e.g. Parvovirus B19) are often associated with a self-limiting symmetrical arthritis of small joints.

Septic polyarthritis caused by direct invasion of the joint by microbes can occur in disseminated staphylococcal and streptococcal infections, gram negative sepsis or bacterial endocarditis. Reactive arthritis, a sterile arthritis mediated by immune mechanisms, is usually seen after genitourinary (Chlamydia) or gastrointestinal (salmonella, shigella, yersinia or campylobacter) infections. It is said that arthritis persisting for more than 6 weeks usually rules out an infective pathology.

Clues from the history and examination:

* Arthritis present for at least 6 weeks before diagnosis (mandatory for diagnosis of JIA).
* Either insidious or abrupt disease onset, often with morning stiffness and arthralgia during the day, joint pain or abnormal joint use, history of school absences or limited ability to participate in physical education classes, spiking fever occurring once or twice each day at about the same time of day all are history findings in children with JIA.
* "How has their general health been?" - Asking about red flags? The presence of systemic symptoms should raise concerns about multisystem illness (e.g. JSLE or inflammatory bowel syndromes and further serious pathology such as malignancy, bacterial infection or trauma (including non-accidental injury; NAI) must be excluded before diagnosing JIA. It is therefore essential to check for the presence of 'red flags Musculoskeletal red flags

Night time wakening with pain Bone pain Fever Anorexia Weight loss Malaise Features suggestive of non-accidental injury

"Did anything precede their symptoms?" - Distinguishing reactive and traumatic causes Typically, reactive arthritis occurs around 7-10 days after the acute illness and spontaneously remits within 2-3 weeks of onset; gastrointestinal infections may cause a reactive arthritis but in the older patient sexually acquired infection needs to be sensitively explored. Falls in children are common and may be a 'red herring' as children with arthritis are often more prone to falling. It is important to explore further for inconsistency or discrepancy between circumstance and degree of injury, which should raise suspicion about NAI.

"What are they like in the morning?"- Mechanical versus inflammatory features.

Joint swelling is a prominent symptom of inflammatory conditions such as JIA, but can be subtle and often missed by parents (as well as health care professionals). To be diagnostic of JIA, joint swelling needs to persist for several weeks (by definition, more than 6 weeks) and other conditions excluded. Morning stiffness may manifest itself through functional change (i.e. difficulty dressing or managing the stairs: "my child walks like an old man") or through a noticeable change in behaviour; parents often mention that their child is particularly miserable in the morning. Prolonged inactivity may precipitate stiffness known as 'gelling', and the child may describe difficulty getting up after sitting for a sustained length of time e.g.

following long car journeys.

"What can they no longer do?" - Developmental milestones

A history of regression of achieved motor milestones is often present with inflammatory joint disease and can manifest as the child becoming 'clumsy' or withdrawing from activity (e.g. no longer walking independently). Regression of a previously attained motor milestone suggests an acquired condition whereas delay alone might suggest a congenital or inherited condition (such as development dysplasia of the hip (DDH) or muscular dystrophy)

- Identifying the cause of polyarthritis may initially look difficult to the uninitiated. However, clinical clues in patient demographics, disease chronology, inflammatory nature, progression, distribution of joint involvement and extra-articular manifestations help narrow the diagnostic possibilities.

Age At the onset of the disease may give clues to the diagnosis. Polyarticular JIA (rheumatoid factor negative), Kawasaki disease (KD) and Henoch Schonlein purpura (HSP) usually present in early childhood. In mid-childhood, juvenile psoriatic arthritis, Juvenile Dermatomyositis (JDMS) and Polyarteritis Nodosa (PAN) have their peak frequencies. Juvenile ankylosing spondylitis (JAS) and SLE typically present in late childhood or early adolescence. Rheumatoid factor positive polyarticular JIA, mimicking the clinical profile of adult RA, usually presents only after the age of 10years.Disorders like gout and crystal deposition disease are extremely uncommon in children.

Sex While many rheumatological disorders (e.g. SLE, polyarticular JIA) have a predilection for girls, there are others (e.g. vasculitides like KD and PAN; Spondyloarthropathies like inflammatory bowel disease and JAS) which are more common in boys.

Onset of Disease and Duration While some arthritides may have an acute onset (e.g. septic arthritis and arthritis associated with KD/HSP) others may have a subacute or chronic insidious course as typically seen in polyarticular chronic insidious course as typically seen in polyarticular JIA or sarcoidosis. Polyarthritis of less than 6 weeks duration is seen in self limiting viral arthritides, rheumatic fever or reactive arthritis. It may sometimes be prudent not to give a label in the first few weeks of the illness when the disease process is still evolving.

Family History Although Mendelian inheritance is not usually seen in inflammatory polyarthritis, familial clustering of cases can be seen in ankylosing spondylitis, inflammatory bowel disease and psoriatic arthritis. The latter condition is especially intriguing because clinical manifestations of psoriasis can be subtle and very variable amongst the family members.

ELIGIBILITY:
Inclusion Criteria:

All patients Attending Rheumatology clinic and unit whom diagnosed as arthritis below the age of 18 years at the onset of presentation who have 1 or more of the following symptoms: swelling or limitation of motion of a joint , morning stiffness and arthralgia during the day, joint pain or abnormal joint use, history of school absences or limited ability to participate in physical education.

Exclusion Criteria:

* Bone or joint trauma
* Hematological disorder (Leukemia, sickle cell disease, thalassemia or hemophilia).
* Patients with chronic diseases (Renal and hepatic diseases).

Ages: 3 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All children below 18 years have arthritis in assiut university children hospital except exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Define prevalence of different types of arthritis in patients attending to assiut university children hospital | Baseline
  Using full history, a clinical examination and investigations can diagnose different types of arthritis attending assiut university children hospital and define prevalence of different types of arthritis